CLINICAL TRIAL: NCT06453525
Title: PrediSuisse: Automatized Assessment of Difficult Airway Using Three Videolaryngoscopes with the Help of Facial Recognition Techniques and Neural Network
Brief Title: PrediSuisse: Automatized Assessment of Difficult Airway
Acronym: PrediSuisse
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Patrick Schoettker, Professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 04062024
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia; Intubation; Difficult or Failed; Airway Complication of Anesthesia
Keywords: Intubation; difficult airway; videolaryngoscopy
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- C-mac: Intubation performed with a C-Mac videolaryngoscope
  Interventions: Other: intubation
- MacGrath: Intubation performed with a MacGrath videolaryngoscope
  Interventions: Other: intubation
- Airtraq: Intubation performed with an Airtraq videolaryngoscope
  Interventions: Other: intubation

INTERVENTIONS:
Other: intubation — Tracheal intubation using one of the three existing videolaryngoscopes

SUMMARY:
In the "PrediSuisse" research project, the investigators aim to create a reliable, reproducible, ultra-portable and radiation-free automatized software, able to identify automatically collected features, facial characteristics, and range of movements, to predict intubation difficulty. The software will generate a difficulty intubation score tailored to three commercially available videolaryngoscopes with different type of blades, corresponding to the predicted endotracheal intubation difficulty while providing the anaesthesiologist a reliable and non-subjective tool to assess individual patient's risks with regards to airway management.

DETAILED DESCRIPTION:
The Swiss multi-institutional research project "PrediSuisse" aims to automatically predict and classify the difficulty of intubation and airway management using three commercially available videolaryngoscopes (VL) by acquiring face/profiles photos and sequences on a training set of 900 patients during the pre-anaesthesia consultation. For each patient, with the help of recently developed Machine Learning (ML), Artificial Intelligence (AI) and Convolutional Neural Network (CNN) techniques, a specially developed software will be trained to provide a predicted airway management difficulty index. This will be performed by correlating those photos/sequences and the real difficulty level of intubation, determined by three experts by reviewing the recordings of the intubations of the training set patients. The software will then be used in routine on a set of 900 other patients to validate the prediction performance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) presenting at the pre-anesthesia consult for an elective general anesthesia necessitating a tracheal intubation
* Signed informed consent.

Exclusion Criteria:

* Patients not speaking French (in Geneva and Lausanne) or Italian (in Lugano).
* Patients previously operated on the airway with anatomical modifications (ENT Flaps, tracheotomies).
* Patients unable to follow procedures or to give consent will also be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years old) presenting at the pre-anesthesia consult for an elective general anesthesia necessitating a tracheal intubation at the University Hospital of Lausanne, Geneva and Cardiocentro Lugano
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Software creation | 18 months
  The primary outcome is to create a reliable, reproducible, ultra-portable and radiation-free automated software, capable of identifying automatically collected features such as facial characteristics, mouth opening, range of motion while moving the neck and thyromental distance to predict intubation difficulty.
  The identification of the difficult intubation score will be compared by the one goven independantly by three airway experts.

SECONDARY OUTCOMES:
Team Communication | 18 months
  The secondary outcome is to evaluate the impact of streaming images of the intubations acquired by the videolaryngoscopy directly to the screens located in the operating room (OR) on communication between healthcare professionals in the OR with the help of a dedicated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- University Hospital Lausanne CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No